CLINICAL TRIAL: NCT03900845
Title: Novel Lower-Limb Prostheses: Comparing Adherence, Perspiration, and Residual Limb Skin Health in a Hot, Humid Environment and During Activities of Daily Living
Brief Title: Adherence and Perspiration While Wearing Lower Limb Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn Klute, Principal Investigator, Seattle Institute for Biomedical and Clinical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-18-1-0559; CDMRP-OR170314 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lower Extremity Amputation
Keywords: lower limb prosthesis; transtibial amputation; below knee amputation; adherence; perspiration

STUDY DESIGN:
Intervention Model Description: This study will use a within-subject crossover design to identify differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort that may exist between the three study prostheses. The three study prostheses include: (1) a perforated elastomeric liner intended to transport perspiration away from the residual limb, (2) a dynamic air exchange - rising edge design (DAE-RED) suspension system expels perspiration to the prosthesis exterior using a hybrid battery-powered pump and a body-weight activated pump that expels perspiration into a distal chamber, and (3) the participant's as-prescribed prosthesis. The order in which participants wear the perforated elastomeric liner and the DAE-RED systems will be randomized (first or third), but the as-prescribed prosthesis will always be worn second.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Environmental Chamber (Experimental): All participants will wear all three study prostheses in an environmental chamber set at 35 degrees Celsius and 50% relative humidity.
  Interventions: Device: Dynamic Air Exchange - Rising Edge Design (DAE-RED); Device: Perforated elastomeric liner; Device: As-prescribed prosthesis
- Field Measurements (Experimental): All participants will wear all three study prostheses in their home, work, and community environments for two weeks.
  Interventions: Device: Dynamic Air Exchange - Rising Edge Design (DAE-RED); Device: Perforated elastomeric liner; Device: As-prescribed prosthesis

INTERVENTIONS:
Device: Dynamic Air Exchange - Rising Edge Design (DAE-RED) — The DAE-RED suspension system expels perspiration to the prosthesis exterior using a hybrid battery-powered pump and a body-weight activated pump. To use the DAE-RED, subjects will be fit with a modified patellar tendon-bearing socket that fits over a custom liner and sock. Up to four air intake ports are located proximally on the liner, approximately 25 mm superior to the socket brim. These ports incorporate a microvalve that allows air to flow into the liner-skin interstitial space while still maintaining a vacuum suspension. Distally, the pin lock has a 3-mm hole along its longitudinal axis that allows perspiration to be expelled into a distal reservoir. The prosthesis will also include: a standard aluminum pylon, pyramid adapters, and an Ossur Proflex XC prosthetic foot with Unity pump and foot cover.
Device: Perforated elastomeric liner — The unique element of this perforated elastomeric liner are small perforations (~0.3 mm diameter), uniformly distributed on a 4 x 5 mm grid, but with no perforations on the distal umbrella, that allow perspiration to be exuded into the liner-socket interstitial space. To use the perforated elastomeric liner, subjects will be fit with a modified patellar tendon-bearing socket that fits over a sock and the perforated elastomeric liner with a pin lock. The sock, worn between the socket and the liner, is used to absorb perspiration that is transported through the perforations in the liner. When needed for residual limb volume control, additional socks will be donned and included in tare weighing. The prosthesis will also include: a standard aluminum pylon, pyramid adapters, and an Ossur Proflex XC prosthetic foot and cosmesis.
  Other Names: Uniprox Softskin Air prosthesis liner
Device: As-prescribed prosthesis — The individual's as-prescribed suspension system is the prosthesis prescription that the patient and their clinical care team believes is the best prosthesis for their needs.

SUMMARY:
Individuals with lower limb amputation often complain about uncomfortable residual limb skin temperatures and the accumulation of sweat inside their prostheses. It doesn't take long before the presence of sweat on the residual limb leads to a lack of confidence in the security of their prosthetic suspension. Some circumstances allow the wearer to doff the prosthesis before it falls off, wipe it and the residual limb dry, and then don it again. Another option is to simply reduce the intensity of activities before sweat becomes a problem. However, the Warfighter amputee may not be afforded such accommodations. For these service personnel, inadequate moisture management can significantly limit or inhibit their mobility. The objective of the proposed research is to provide lower limb amputees who work in demanding environments with a prosthesis that remains secure despite profuse residual limb sweating without compromising residual limb health and comfort.

The aim of this research is to compare three different, lower limb prosthetic suspension systems and identify which is most effective at maintaining a secure adherence when worn in conditions that result in profuse sweating. The investigators also aim to compare how the three study prostheses effect residual limb skin health and comfort when participants pursue their usual activities in the home, work, and community environments.

To achieve these aims, the investigators will to recruit 25 below-knee amputees. Each subject will be asked to be asked to wear: (1) their as-prescribed prosthesis, (2) a prosthesis with a perforated elastomeric liner that allows sweat to flow away from the skin, and (3) a prosthesis that has a battery and body-weight activated pump to flow air between the prosthesis and the residual limb skin, allowing expulsion of any accumulated sweat. Subjects will wear each of these prostheses in the home, work, and community environments for two weeks, after which the investigators will measure their residual limb health and comfort. Subjects will then walk on a treadmill in a room whose climate will be set to Middle East-like conditions: 35 °C (95 °F) and 50% relative humidity. After 30 minutes, the investigators will measure any slippage of their prosthesis relative to their limb and how much sweat is expelled. The investigators hypothesize there will be differences in the amount of slippage, residual limb health, and comfort between the three prostheses.

DETAILED DESCRIPTION:
Individuals with lower limb amputation often complain about uncomfortable residual limb skin temperatures, accumulation of perspiration inside their prostheses, and loss of confidence in suspension security that often leads them to cease their activities or, in demanding circumstances, may lead to their prosthesis falling off. Most amputees can sense the impending loss of suspension during vigorous activities and can stop, doff the prosthesis, wipe it and the residual limb dry, and then don it again. However, the Warfighter amputee may not be afforded such accommodations.

The investigators will compare the performance of an individual's as-prescribed suspension with two exciting alternatives: a new-to-market liner intended to transport perspiration away from the skin and an improved version of the Dynamic Air Exchange (DAE) suspension system the investigators developed. The new-to-market suspension system consists of a perforated elastomeric liner that allows perspiration to be exuded into the liner-prosthesis space. Anecdotal reports suggest this liner (Uniprox's SoftSkin Air), can maintain suspension during profuse perspiration, but may result in excessive skin dryness and discomfort. The improved Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension expels accumulated perspiration using a vacuum pump like its predecessor, but incorporates hybrid, body-weight activated pump to minimize battery consumption and a revised ventilation system obviating the need for undesirable exterior tube connections.

The objective of the proposed research is to provide lower limb amputees who work in demanding environments with a prosthesis that remains secure despite profuse residual limb perspiration without compromising residual limb health and comfort.

The proposed research has two specific aims: (1) compare three different, lower limb prosthetic suspension systems and identify which is most effective at maintaining a secure adherence when worn in conditions that result in profuse perspiration, and (2) compare how the three suspension systems effect residual limb skin health and comfort when participants pursue their usual activities in the home, work, and community environments.

The investigators will recruit unilateral transtibial amputees who are successful ambulators on their as-prescribed prosthesis and collect baseline data (residual limb skin hydration, transepidermal water loss (skin barrier function), and Socket Comfort Score). After fitting the participants with Uniprox and DAE-RED prostheses, subjects will wear one of these study prostheses (random order) for two weeks, after which the investigators will measure their skin hydration, transepidermal water loss, and Socket Comfort Score. The subject will then enter our environmental chamber (35° C and 50% relative humidity) and sit for a 30-minute acclimation period. The subject will then walk for 30 minutes on a treadmill at their self-selected speed. Subjects will then exit the environmental chamber and sit for 30 minutes in a comfortable climate (~20° C and 50% relative humidity). The amount of slippage, along with the perspiration accumulated/expelled, will be then be measured. Subjects will then be fit with their as-prescribed prosthesis and the protocol repeated to washout intervention effects. Finally, subjects will be fit with the other study prosthesis (either Uniprox or DAE-RED) and repeat the protocol.

After wearing the prostheses in our environmental chamber set to Middle East-like conditions (35 °C and 50% relative humidity), the investigators hypothesize:

H1.1 The amount of slippage (loss of adherence) will be different between the three suspension systems.

H1.2 The amount of perspiration expelled will be different between the Uniprox and DAE-RED.

After wearing the study prostheses in the home, work, and community environments for two weeks, the investigators hypothesize:

H2.1 Residual limb skin hydration will be different between the three suspension systems.

H2.2 Residual limb transepidermal water loss will be different between the three suspension systems.

H2.3 The Socket Comfort Score will be different between the three suspension systems.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Been fit with a prosthesis and used it for at least six months
* Wear the prosthesis for four or more ours on an average day
* Ambulate without upper extremity aids
* Able to walk for 30 minutes on a treadmill

Exclusion Criteria:

* Improper fit and suspension with current prosthesis and one cannot be achieved with clinical resources (determined at initial visit)
* Current skin irritation or injury on residual limb
* Osteoarthritis, injury, or pain that interferes with walking ability
* Currently incarcerated
* Pregnant (determined via self-report)
* Inadequate cognitive function or language proficiency to consent to participate
* High (>20%) coronary heart disease risk at 10 years as determined by heir Framingham Risk Score

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — Dept. of Veterans Affairs
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset in machine-readable format will be created and shared for all individual participant data (IPD) that underlie results in a publication. The investigators will follow 164.514(a) of the HIPAA Privacy Rule for de-identification of IPD.
Time Frame: Within six months after publication of final study findings.
Access Criteria: Open access through Pubmed Central, SimTk, PhysioNet, or other similar open-source data repository websites. The investigators will work with manuscript publishers when possible to link the final study data sets to an appendix or supplemental materials on the publisher websites.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants was performed at a US Veterans Hospital.
Pre-assignment Details: Twenty eligible individuals (17 male, 3 female) were enrolled in the study. All considered themselves moderately active community ambulators. Twelve individuals terminated before randomization: one withdrew due to health issues, one did not feel strong enough to complete the protocol, one left the country, five had prosthetic fitting issues, and four were lost to follow up after consent.
Groups:
- PERF, Then RX, Then DAE-RED: A within-subject crossover experiment was conducted to determine if differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort exist between three study suspension systems. The three suspension systems included: (1) a perforated elastomeric liner (PERF) liner intended to transport perspiration away from the residual limb, (2) a Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension system that expels perspiration to the prosthesis exterior using a hybrid battery and body weight actuated vacuum pumps, and (3) the participant's as-prescribed (RX) prosthesis. The order in which participants wore the PERF and DAE-RED systems was randomized (first or third), but the RX prosthesis was always worn second.
  This study was conducted over 6 weeks. Subjects were fit with the study prostheses (PERF and DAE-RED) and then randomized to first wear either the PERF or DAE-RED prosthesis for two weeks before returning for data collection. Subjects were then fit with their RX prosthesis which they wore for the next two weeks to wash out intervention effects before returning for data collection. Subjects were then fit with the remaining study prosthesis (either the PERF or DAE-RED) which they wore for two weeks before returning for data collection. After wearing all three prostheses, the protocol was complete.
  Participants in this group first wore PERF for two weeks, then RX for two weeks, and then DAE-RED for two weeks.
- DAE-RED, Then RX, Then PERF: A within-subject crossover experiment was conducted to determine if differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort exist between three study suspension systems. The three suspension systems included: (1) a perforated elastomeric liner (PERF) liner intended to transport perspiration away from the residual limb, (2) a Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension system that expels perspiration to the prosthesis exterior using a hybrid battery and body weight actuated vacuum pumps, and (3) the participant's as-prescribed (RX) prosthesis. The order in which participants wore the PERF and DAE-RED systems was randomized (first or third), but the RX prosthesis was always worn second.
  This study was conducted over 6 weeks. Subjects were fit with the study prostheses (PERF and DAE-RED) and then randomized to first wear either the PERF or DAE-RED prosthesis for two weeks before returning for data collection. Subjects were then fit with their RX prosthesis which they wore for the next two weeks to wash out intervention effects before returning for data collection. Subjects were then fit with the remaining study prosthesis (either the PERF or DAE-RED) which they wore for two weeks before returning for data collection. After wearing all three prostheses, the protocol was complete.
  Participants in this group first wore DAE-RED for two weeks, then RX for two weeks, and then PERF for two weeks.
Period: First Intervention (2 weeks)
Arm/Group | PERF, Then RX, Then DAE-RED | DAE-RED, Then RX, Then PERF
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0
Period: Second Intervention (2 weeks)
Arm/Group | PERF, Then RX, Then DAE-RED | DAE-RED, Then RX, Then PERF
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0
Period: Third Intervention (2 weeks)
Arm/Group | PERF, Then RX, Then DAE-RED | DAE-RED, Then RX, Then PERF
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Individuals With Unilateral Transtibial Amputation: A within-subject crossover experiment was conducted to determine if differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort exist between three study suspension systems. The three suspension systems included: (1) a perforated elastomeric liner (PERF) liner intended to transport perspiration away from the residual limb, (2) a Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension system that expels perspiration to the prosthesis exterior using a hybrid battery and body weight actuated vacuum pumps, and (3) the participant's as-prescribed (RX) prosthesis. The order in which participants wore the PERF and DAE-RED systems was randomized (first or third), but the RX prosthesis was always worn second.
Arm/Group | Individuals With Unilateral Transtibial Amputation
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: The amount of slippage (loss of adherence) will be determined by measuring the distance between a mark on the skin and the proximal border of the liner. Adherence will be measured in millimeters.
Time Frame: After the 90-minute rest-walk-rest protocol where subjects enter our environmental chamber for a 30-minute seated acclimation and a 30-minute treadmill walk and then exit the chamber for a 30-minute seated rest.
Measure: Mean (Standard Error); unit: millimeters
Groups:
- As-Prescribed (RX): The individual's as-prescribed suspension system is the prosthesis prescription that the patient and their clinical care team believes is the best prosthesis for their needs.
- Perforated Liner (PERF): The unique element of the PERF are small perforations (~0.3 mm diameter), uniformly distributed on a 4 x 5 mm grid, but with no perforations on the distal umbrella, that allow perspiration to be exuded into the liner-socket interstitial space. To use the perforated elastomeric liner, subjects will be fit with a modified patellar tendon-bearing socket that fits over a sock and the perforated elastomeric liner with a pin lock. The sock, worn between the socket and the liner, is used to absorb perspiration that is transported through the perforations in the liner. When needed for residual limb volume control, additional socks will be donned and included in tare weighing. The prosthesis will also include: a standard aluminum pylon, pyramid adapters, and an Ossur Proflex XC prosthetic foot and cosmesis.
Arm/Group | Dynamic Air Exchange - Rising Edge Design (DAE-RED) | As-Prescribed (RX) | Perforated Liner (PERF)
Number analyzed (Participants) | 8 | 8 | 8
millimeters | 1 (1) | 8 (4) | 3 (2)
Statistical Analysis 1: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs As-Prescribed (RX) vs Perforated Liner (PERF); Hypothesis testing for the association between outcome and study interventions was carried out using conditional F-tests; Test type: Superiority; p = .037, Regression, Linear
Statistical Analysis 2: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs As-Prescribed (RX); Test type: Superiority; p = 0.031, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method
Statistical Analysis 3: Comparison: As-Prescribed (RX) vs Perforated Liner (PERF); Test type: Superiority; p = 0.220, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method
Statistical Analysis 4: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs Perforated Liner (PERF); Test type: Superiority; p = 0.510, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method

2. Primary Outcome: Expelled Perspiration
Description: The amount of expelled perspiration will be determined by tare weight. Expelled perspiration will be measured in grams.
Time Frame: as for outcome 1
Population: The As-Prescribed (RX) prosthesis cannot expel perspiration. No measurements were performed on this group.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Dynamic Air Exchange - Rising Edge Design (DAE-RED) | As-Prescribed (RX) | Perforated Liner (PERF)
Number analyzed (Participants) | 8 | 0 | 8
grams | 0.1 (0.01) |  | 0.2 (0.1)
Statistical Analysis 1: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs Perforated Liner (PERF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.380, Regression, Linear

3. Secondary Outcome: Skin Hydration
Description: Skin hydration will be measured with a specialized instrument (Corneometer). A probe, acting as a capacitor, will apply an electric field to penetrate the skin (i.e., epidermis stratum corneum) on the posterior compartment of the residual limb to a depth of 10 to 20 μm. The amount of electrical charge stored by the capacitor is a function of skin hydration. Greater water content is proportional to higher capacitance, which is converted to converted to arbitrary units from 0 to 99. Skin hydration of less than 30 au is an indicator of very dry skin while greater than 40 au indicates sufficiently moisturized skin.
Time Frame: After wearing the study prosthesis in the home, work, and community environments for two weeks
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Dynamic Air Exchange - Rising Edge Design (DAE-RED) | As-Prescribed (RX) | Perforated Liner (PERF)
Number analyzed (Participants) | 8 | 8 | 8
Units on a scale | 18 (4) | 21 (4) | 26 (4)
Statistical Analysis 1: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs As-Prescribed (RX) vs Perforated Liner (PERF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.160, Regression, Linear

4. Secondary Outcome: Transepidermal Water Loss
Description: Transepidermal water loss will be measured with a specialized instrument (Tewameter). A hollow cylinder probe with two pairs of sensors (temperature and relative humidity) will measure the density gradient of the water evaporation on the posterior compartment of the residual limb in units of g/m2/h. Transepidermal water loss between 10 and 15 g/h/m2 is an indicator of healthy skin. Transepidermal water loss of less than 10 g/h/m2 indicates very healthy skin.
Time Frame: After wearing the study prosthesis in the home, work, and community environments for two weeks
Measure: Mean (Standard Error); unit: grams per hour per square meter
Arm/Group | Dynamic Air Exchange - Rising Edge Design (DAE-RED) | As-Prescribed (RX) | Perforated Liner (PERF)
Number analyzed (Participants) | 8 | 8 | 8
grams per hour per square meter | 12.3 (2.2) | 12.8 (2.2) | 9.3 (2.2)
Statistical Analysis 1: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs As-Prescribed (RX) vs Perforated Liner (PERF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.400, Regression, Linear

5. Secondary Outcome: Satisfaction With the Prosthesis
Description: An 11-point Likert scale will be used to record the subject's perception of satisfaction with the study prostheses. Participants will be asked to rate their satisfaction with the prosthesis on a 0 - 10 scale where 0 and 10 represent the least amount of satisfaction and the most amount of satisfaction imaginable, respectively. A higher score indicates a better outcome.
Time Frame: After wearing the study prosthesis in the home, work, and community environments for two weeks
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Dynamic Air Exchange - Rising Edge Design (DAE-RED) | As-Prescribed (RX) | Perforated Liner (PERF)
Number analyzed (Participants) | 8 | 8 | 8
Units on a scale | 7 (1) | 8 (1) | 7 (1)
Statistical Analysis 1: Comparison: Dynamic Air Exchange - Rising Edge Design (DAE-RED) vs As-Prescribed (RX) vs Perforated Liner (PERF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.320, Regression, Linear

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- PERF, Then RX, Then DAE-RED: A within-subject crossover experiment was conducted to determine if differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort exist between three study suspension systems. The three suspension systems included: (1) a perforated elastomeric liner (PERF) liner intended to transport perspiration away from the residual limb, (2) a Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension system that expels perspiration to the prosthesis exterior using a hybrid battery and body weight actuated vacuum pumps, and (3) the participant's as-prescribed (RX) prosthesis. The order in which participants wore the PERF and DAE-RED systems was randomized (first or third), but the RX prosthesis was always worn second.
  Participants in this group first wore PERF for two weeks, then RX for two weeks, and then DAE-RED for two weeks.
- DAE-RED, Then RX, Then PERF: A within-subject crossover experiment was conducted to determine if differences in adherence (slippage), expulsion of perspiration, residual limb health, and comfort exist between three study suspension systems. The three suspension systems included: (1) a perforated elastomeric liner (PERF) liner intended to transport perspiration away from the residual limb, (2) a Dynamic Air Exchange - Rising Edge Design (DAE-RED) suspension system that expels perspiration to the prosthesis exterior using a hybrid battery and body weight actuated vacuum pumps, and (3) the participant's as-prescribed (RX) prosthesis. The order in which participants wore the PERF and DAE-RED systems was randomized (first or third), but the RX prosthesis was always worn second.
  Participants in this group first wore DAE-RED for two weeks, then RX for two weeks, and then PERF for two weeks.
Arm/Group | PERF, Then RX, Then DAE-RED | DAE-RED, Then RX, Then PERF
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03900845/Prot_003.pdf
  • Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03900845/SAP_001.pdf
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03900845/ICF_002.pdf